CLINICAL TRIAL: NCT04675502
Title: Comparison of the Effects of a Supervised Exercise Program and a Home Exercise Program in Patients With Systemic Sclerosis
Brief Title: Effects of a Supervised Exercise Program and a Home Exercise Program in Patients With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hazal Yakut, Principal investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3701-GOA
Record Dates: First submitted 2020-11-25; First posted 2020-12-19 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-02

CONDITIONS: Systemic Sclerosis; Home Exercise; Aerobic Exercise
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise Group (Experimental): Exercise programs including warm-up, loading, cooling, and relaxation exercises are shown. The warm-up period is consist of light-paced walking, active movements of several large muscle groups. In this loading program; respiratory control training, breathing exercises, posture exercises with respiratory control , walking on the treadmill for 20 minutes without inclination , pedaling in the bicycle ergometer for 10 minutes is taken. Stretching exercises are done during the cooling period. This group was included in an exercise program 2 days a week, 45-90 minutes, for 12 weeks, accompanied by a specialist physiotherapist to the pulmonary rehabilitation unit in the chest diseases ward.
  Interventions: Other: supervised Exercise training
- Home Exercise Group (Experimental): For patients to do at home (respiratory control training, shrunken lip breathing exhaustion, diaphragmatic, thoracic expansion exercises, posture exercises with respiratory control (pectoral stretching, four-way trunk exercises, head and neck exercises, bilateral shoulder flexion and abduction exercises), sitting and standing exhaustion, and brisk walking to reach 60-85% of the person's maximum heart rate.)), exercises is taught. Patients were asked to do the exercises at home for 45-90 minutes, 2 days a week, for 12 weeks. Participants of the control group are contacted every two weeks via communication methods such as e-mail, message and telephone conversation.Exercise diary is given to all patients and is taken from them at the end of the study.
  Interventions: Other: home exercise trainig

INTERVENTIONS:
Other: supervised Exercise training — warm-up, loading (respiratory control training, breathing exercises, posture exercises with respiratory control , walking on the treadmill for 20 minutes without inclination , pedaling in the bicycle ergometer for 10 minutes), cooling, and relaxation exercises
  Arms: Supervised Exercise Group
Other: home exercise trainig — Warm-up, loading (respiratory control training, shrunken lip breathing exhaustion, diaphragmatic, thoracic expansion exercises, posture exercises with respiratory control (pectoral stretching, four-way trunk exercises, head and neck exercises, bilateral shoulder flexion and abduction exercises), cooling and relaxation exercises
  Arms: Home Exercise Group

SUMMARY:
Scleroderma, also called systemic sclerosis (SSc); It is a heterogeneous multiorgan disease of unknown etiology characterized by vasculopathy, autoimmunity and fibrous tissue. It is stated in studies that cardiac and pulmonary systems are affected in patients with SSc and these effects affect the aerobic capacity, physical functions and quality of life of patients negatively by disrupting their pulmonary and musculoskeletal functions. However, considering the treatment approaches in scleroderma patients, the number of studies evaluating the effectiveness of pulmonary rehabilitation and exercises is limited. Therefore, the purpose of our study; Comparison of the effects of a supervised exercise program and a home exercise program in patients with Systemic Sclerosis.

DETAILED DESCRIPTION:
Cases are divided into two groups as supervised exercise and home exercise program by closed envelope randomization method. All patients are informed about risk factors and risk factor management. All patients are trained 3 days in the first week under the supervision of a physiotherapist to learn individual exercise programs. Supervised exercise programs including warm-up, loading, cooling, and relaxation exercises are shown. The warm-up period is consist of light-paced walking, active movements of several large muscle groups. During the loading period respiratory control training, breathing exercises (Shrunken lip breathing exhaustion, diaphragmatic, thoracic expansion exercises), posture exercises with respiratory control (pectoral stretching, four-way trunk exercises, head-neck exercises, bilateral shoulder flexion and abduction exercises, sitting on a chair, standing up exercise. ), walking on the treadmill for 5-15 minutes without inclination and at a constant speed, starting with 3 minutes without load, continuing with a load of 20 watts and 3 minutes, and reaching a submaximal load with 3 watt increments every 10 seconds, pedaling in the bicycle ergometer is taken. Stretching exercises are done during the cooling period. This group was included in an exercise program 2 days a week, 45-90 minutes, for 12 weeks, accompanied by a specialist physiotherapist in the pulmonary rehabilitation unit in the chest diseases ward. The same exercises (respiratory control training, shrunken lip breathing exhaustion, diaphragmatic, thoracic expansion exercises, posture exercises with respiratory control (pectoral stretching, four-way trunk exercises, head and neck exercises, bilateral shoulder flexion and abduction exercises), sitting and standing exhaustion, and brisk walking to reach 60-85% of the person's maximum heart rate.)) were taught to the home exercise group and given in the form of a brochure and they were asked to do these exercises at home 2 days a week for 12 weeks. Participants of the home exercise group are contacted every two weeks via communication methods such as e-mail, message and telephone conversation. Exercise diary is given to all patients and is taken from them at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Stable clinical status for at least two weeks
* Walking independently
* Volunteer for research study

Exclusion Criteria:

* Having unstable angina
* Having uncontrolled hypertension
* Having hemodynamic instability
* Participating in any exercise program in the last six months
* Having a major orthopedic or neurological problem that limits functionality

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity | Baseline, 12th week
  Pulmonary function test was applied by Sensor Medics Vmax 22 0,6-2B version spirometer (ERS 1993 Uptake + Zapleta, SensorMedics, Inc, Anaheim, CA, USA). Forced vital capacity (FVC) percent was recorded according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria
Change in Forced Expiratory Volume in One Second | Baseline, 12th week
  Pulmonary function test was applied by Sensor Medics Vmax 22 0,6-2B version spirometer (ERS 1993 Uptake + Zapleta, SensorMedics, Inc, Anaheim, CA, USA). Forced expiratory volume in one second (FEV1) percent was recorded according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria
Change in Forced expiratory volume in one second / Forced vital capacity | Baseline, 12th week
  Pulmonary function test was applied by Sensor Medics Vmax 22 0,6-2B version spirometer (ERS 1993 Uptake + Zapleta, SensorMedics, Inc, Anaheim, CA, USA). Forced expiratory volume in one second (FEV1)/Forced vital capacity (FVC) ratio percent was recorded according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria
Change in diffusion capacity | Baseline, 12th week
  Single breath carbon monoxide method was used in diffusion capacity for carbon monoxide (DLCO) percent measurement
Change in Maximal Expiratory Pressure | Baseline, 12th week
  Electronic mouth pressure measuring device was used for respiratory muscle strength. Maximal expiratory pressure (MEP) was measured. MEP was measured from total lung capacity performing a maximal expiratory effort against an occluded airway. MEP measurements was repeated three times, and the maximum percent achieved was recorded
Change in Maximal Inspiratory Pressure | Baseline, 12th week
  Electronic mouth pressure measuring device was used for respiratory muscle strength. Maximal inspiratory pressure (MIP) was measured. MIP was measured from residual volume upon a maximal inspiratory effort against an occluded airway. occluded airway. MIP measurements was repeated three times, and the maximum percent achieved was recorded.
Change in functional capacity | Baseline, 12th week
  Six-minute walk test (6MWT) is a valid, reliable and useful test for assessing functional capacity of patients. This test assesses distance walked over 6 minutes as a sub maximal test of aerobic capacity/endurance.
Change in peripheral muscle strength | Baseline, 12th week
  The Jamar Handgrip Dynamometer is an instrument for measuring the maximum isometric strength of the hand and forearm muscles. Quadriceps isometric muscle strength is measured with a Hand Held Dynamometer.

SECONDARY OUTCOMES:
Change in severity of dyspnoea | Baseline, 12th week
  Modified Medical Research Council (mMRC) dyspnea scale is a valid and reliable test for measuring the severity of dyspnea. This scale ranges from 0 to 4. A higher value represents a worse outcome
Change in fatigue | Baseline, 12th week
  The Fatigue Impact Scale that questions how much fatigue the scale has experienced in a month, taking as a reference a total of 40 items, including the day of application. Scores between 0 and 4 points are given for each item, and the maximum score is calculated to be 160.High score indicates a high level of fatigue.
Change in quality of life:Health Assessment Questionnaire Disability Index | Baseline, 12th week
  Health Assessment Questionnaire Disability Index (HAQ-DI) measures disability, function and quality of life with 8 functional domains of physical capacity (dress / get up / eat / walk / hygiene / to reach objects / grip / activities) which consists of 20 items. Each item scored between 0 (without any difficulty) and 3 (unable to do). The scale is scored between 0 and 60 and the high score indicates poor health quality status
Change in quality of life: Scleroderma Health Assessment Questionnaire | Baseline, 12th week
  The Scleroderma Health Assessment Questionnaire (SHAQ)-global score which was calculated by adding five SSc-related VAS to eight HAQ-DI domains and dividing the sum by 13. he subscales are scored between 0 and 3 and the high score indicates poor health status
Change in quality of life: Short Form-36 Quality of Life Questionnaire | Baseline, 12th week
  SF-36 measures health-related quality of life and consists of 36 items in total and includes two subscales that are physical and mental. The subscales are scored between 0 and 100 and the low score indicates poor health status

CONTACTS AND LOCATIONS:
Overall Officials: Hazal Yakut, PT,MSc, Principal Investigator — Dokuz Eylul University; Sevgi Özalevli, PT,PhD, Study Director — Dokuz Eylul University; Gerçek Can, MD, Study Chair — Dokuz Eylul University; Aylin Özgen Alpaydın, MD, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylül Üniversitesi School of Physical Therapy and Rehabilitation, Izmir, İzmir, Turkey, Turkey (Türkiye)